CLINICAL TRIAL: NCT05531175
Title: INVESTIGATION OF THE EFFECT OF REIKI APPLICATION ON PAIN, FATIGUE AND ITCHING IN HEMODIALYSIS PATIENTS
Brief Title: REIKI APPLICATION PAIN, FATIGUE AND ITCHING IN HEMODIALYSIS PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Esra Baser Akin, Research Asisstant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-06/24
Record Dates: First submitted 2022-08-27; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): A total of 10 sessions of reiki were applied to the patients in the intervention group twice a week for 5 weeks, lasting 40-45 minutes during dialysis. The scales were administered to the individuals in the intervention groups three times in total.
  Interventions: Other: Reiki apply
- Control Group (No Intervention): No treatment was applied to the control group. The scales were administered to the individuals in the control groups three times in total.

INTERVENTIONS:
Other: Reiki apply — The intervention group is the group in which reiki is applied. They receives 3 sessions of hemodialysis per week.
  Arms: İntervention Group

SUMMARY:
The research sample consisted of 74 individuals, including the intervention group (n=37) and the control group (n=37), who received hemodialysis treatment at Sivas Cumhuriyet University Application and Research Hospital Hemodialysis Unit, Sivas Numune Hospital Hemodialysis Unit and Private ONR Dialysis Center. The data of the study were collected using the Patient Description Form, the Patient Clinical Parameters Form (Some Treatment Data and Laboratory Results, Measurement of Pain Intensity), Visual Analogue Scale (VAS), McGill Melzack Pain Questionnaire, Piper Fatigue Scale, and 5-D Itch Scale. A total of 10 sessions of reiki were applied to the patients in the intervention group twice a week for 5 weeks, lasting 40-45 minutes during dialysis. No treatment was applied to the control group. The scales were administered to the individuals in the intervention and control groups three times in total.

ELIGIBILITY:
Inclusion Criteria:

* The research sample consisted of patients who had no difficulties in communicating and had no mental problems, who had undergone hemodialysis treatment for at least one year, who were 18 years of age or older and who agreed to participate in the study, who did not receive complementary alternative treatment for symptom management, and who experienced symptoms of fatigue, itching and pain.

Exclusion Criteria:

* Those younger than 18 years of age, those receiving hemodialysis treatment for less than a year, those with communication difficulties, those with psychiatric problems, and those who wanted to leave the study were not included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-05-22 (Actual)

PRIMARY OUTCOMES:
Pain Status Visual Analog Scale Visual analog scale and A short form of the McGill Pain Questionnaire | Pain assessment was made at the first interview (basaline), in the second week of the reiki application, and in the fifth week of the reiki application. Changes in the pain level of the patients were observed.
  It is a scale used to evaluate the pain experienced by patients. It is a scale used to evaluate the pain experienced by patients. Hastaların yaşadığı ağrıyı değerlendirmek için kullanılan bir ölçektir. It is a scale that is used to evaluate the pain experienced by patients. Hastaların yaşadığı ağrıyı değerlendirmek için kullanılan bir ölçektir. Scale; It contains the numbers "starting 0 (no pain)" and "10 (severe pain)" at the other end.
Pain Status A short form of the McGill Pain Questionnaire Visual analog scale and A short form of the McGill Pain Questionnaire | Pain assessment was made at the first interview (basaline), in the second week of the reiki application, and in the fifth week of the reiki application. Changes in the pain level of the patients were observed.
  The McGill Melzack Pain Questionnaire (MASF) was developed in 1971 by Melzack and Targerson. It consists of three parts evaluating pain pattern, current pain index, and pain scale score.
Piper Fatigue Scale | Fatigue assessment was made at the first interview (basaline), in the second week of the reiki application, and in the fifth week of the reiki application. Changes in the fatigue level of the patients were observed.
  The scale was developed by Piper et al. in 1998. The scale, which subjectively evaluates the patient's fatigue in four dimensions, consists of 27 items in total. The sub-dimensions of the scale, the behavior/violence sub-dimension (2-7 items); affect sub-dimension (items 8-12), which includes the emotional meaning of fatigue; it is the sensory sub-dimension (13-17 items) showing the physical, psychological and emotional symptoms of fatigue, and the cognitive/spiritual sub-dimension (18-23 items) showing the effect of fatigue on cognitive and mental state. The total score is obtained by adding each item and dividing it by the number of items.
5-D Itch Scale | Itching assessment was made at the first interview (basaline), in the second week of the reiki application, and in the fifth week of the reiki application. Changes in the itching level of the patients were observed.
  The 5-D Itch Scale was developed by Elman, Hyman, Gabriel and Mayo in 2010. The scale consists of 5 dimensions and 8 variables as the duration, severity, course of itching, the area of restriction in activities of daily living and its distribution in the body. The scale is scored between a minimum of 5 (no itching) and a maximum of 25 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra BAŞER AKIN, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
PhD thesis submission exam
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 22 September 2022

REFERENCES:
- [Derived] Baser Akin E, Mollaoglu M. Investigation of the Effect of Reiki on Pain, Fatigue, and Itching in Hemodialysis Patients: Randomized Controlled Trial. Hemodial Int. 2025 Apr;29(2):201-213. doi: 10.1111/hdi.13203. Epub 2025 Feb 5. PMID 39908578